CLINICAL TRIAL: NCT06982274
Title: Combination of Oral Arsenic With ATRA and Minimal-Dose Chemotherapy for Newly Diagnosed Patients With Acute Promyelocytic Leukemia: a Study by the International Consortium on APL
Brief Title: Oral Arsenic With ATRA for Newly Diagnosed Patients With Acute Promyelocytic Leukemia
Acronym: IC-APL2020
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: American Society of Hematology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1483/2019
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Acute Promyelocytic Leukemia (APL)
Keywords: Acute promyelocytic leukemia; Oral arsenic; Survival; All trans-retinoic acid
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Arsenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proposed protocol (Experimental): Oral Arsenic + ATRA with low-dose daunorubicin for high-risk patients
  Interventions: Drug: Realgar-Indigo Naturalis Formulation

INTERVENTIONS:
Drug: Realgar-Indigo Naturalis Formulation — Oral Arsenic (Realgar-Indigo Naturalis Formulation) plus ATRA for low-intermediate risk APL pts, combined with daunorubicin for high-risk during induction
  Other Names: Oral Arsenic

SUMMARY:
It is a non-randomized, multicenter, prospective study, aiming to treat patients with newly diagnosed acute promyelocytic leukemia with a combination of oral arsenic and atra, with low dose chemotherapy for those with high-risk disease (white blood cell count above 10x10a9/L). The primary objective is to assess the 2-year overall survival (OS) in these patients, comparing with the historical control group of patients treated with ATRA/chemotherapy according to the IC-APL 2006 protocol.

DETAILED DESCRIPTION:
This is a non-randomized, multicenter, prospective study aimed at treating patients with newly diagnosed acute promyelocytic leukemia (APL) using a combination of oral arsenic and ATRA. For patients classified as high-risk (white blood cell count >10×10⁹/L), low-dose chemotherapy will be added. The primary objective is to evaluate the 2-year overall survival (OS) in these patients, comparing it to a historical control group treated with ATRA and chemotherapy according to the IC-APL 2006 protocol. Secondary objectives include: Comparing complete response rates, disease-free survival, cumulative incidence of relapse, and early mortality with those reported in the IC-APL 2006 study (historical controls), as well as with outcomes reported in developed countries; Comparing the cumulative incidence of myelodysplasia or secondary leukemia; Comparing the toxicity profile with historical data; Assessing the molecular remission rate after consolidation; Evaluating the reduction in PML/RARA transcript levels during treatment; Comparing the duration of patient hospitalization with historical results.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* New diagnosis of APL by cytomorphology, confirmed for molecular analysis
* Age ≥18 and ≤75 years
* Serum total bilirubin ≤ 3.0 mg/dl (≤ 51 μmol/l)
* Serum creatinine ≤ 3.0 mg/dl (≤ 260 μmol/l)
* Women must meet at least one of the following criteria to be eligible for inclusion in the study: Postmenopausal (12 months of amenorrhea or 6 months of amenorrhea with serum FSH > 40 U/ml); After undergoing hysterectomy or bilateral oophorectomy; Continuous and correct use of a contraceptive method with a Pearl Index <1% (e.g., implants, oral contraceptives, intrauterine devices); Sexual abstinence; Vasectomy of sexual partner.

Exclusion Criteria:

* High-risk patients who are not eligible for chemotherapy according to the judgment of the treating physician;
* Age <18 or >75 years
* Other active malignancy at the time of study entry
* Lack of diagnostic confirmation at the genetic level
* Significant arrhythmias, ECG abnormalities, or neuropathy: Congenital long QT syndrome; History or presence of significant ventricular or atrial tachyarrhythmia; Clinically significant resting bradycardia (<50 beats per minute); QTc > 500 ms on ECG screening for both sexes; Right bundle branch block with left anterior hemiblock or bifascicular block
* High-risk patients with other cardiac contraindications for intensive chemotherapy (LVEF < 50%)
* Uncontrolled and potentially fatal infections
* Severe uncontrolled pulmonary or cardiac disease
* Severe hepatic or renal dysfunction
* Known HIV and/or hepatitis C infection
* Pregnant or breastfeeding women
* Allergy to the study drug or excipients in the study medication
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or the assessment of study outcomes
* Use of other investigational drugs at the time of enrollment or within 30 days before study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2 years
  This endpoint includes death from any cause, including early death, death due to disease progression, or any death occurring after achieving complete remission.

SECONDARY OUTCOMES:
Complete hematologic response rate after induction. | 30 days
  Absence of leukemic promyelocytes in the peripheral blood and bone marrow (<5% blasts), recovery of normal blood counts (ANC ≥ 1.0 × 10⁹/L and platelets ≥ 100 × 10⁹/L), no extramedullary disease, and resolution of coagulopathy.
Early death rate during induction | 30 days
  Death before blood cell counts recovery during induction.
Disease-free survival rate | 2 years
  The proportion of patients who remain alive and in complete remission, without evidence of relapse, for at least two years following achievement of initial complete remission.
Cumulative incidence of myelodysplasia and secondary leukemia | 5 years
  The proportion of patients who develop myelodysplastic syndromes or secondary leukemia after treatment.
Cumulative incidence of relapse | 2 years
  The proportion of patients who experience a relapse of acute leukemia within two years of achieving complete remission, accounting for competing risk of death without relapse.
Molecular remission rate after consolidation | 150 days
  The proportion of patients who achieve a negative molecular test by PCR for PML-RARA after completing the consolidation phase of treatment.
PML/RARA transcript level during treatment | Each 3 months
  The quantitative measurement of the PML/RARA fusion gene transcript, assessed by PCR, at various stages of therapy.
Days of hospitalization during treatment | 180 days
  The total length of time a patient spends in the hospital for the administration of treatment, management of complications, or observation during the course of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo M Rego, MD PhD, Principal Investigator — Instituto do Cancer do Estado de Sao Paulo
Locations (1):
- Instituto do Cancer do Estado de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva WF, Kim HT, Undurraga MS, Navarro-Cabrera JR, Salinas V, Muxi P, Melo RAM, Gloria ABF, Pagnano KBB, Nunes EC, Bittencourt RI, Rojas N, Truyenque SMQ, Ayala-Lugo AI, Oliver AC, Figueiredo-Pontes LL, Traina F, Moreira F, Fagundes EM, Duarte BKL, Mora-Alferez AP, Ortiz P, Untama JL, Tallman MS, Ribeiro RC, Ganser A, Dillon RJ, Valk PJM, Sanz MA, Lowenberg B, Berliner N, Rego EM. Early death and intracranial hemorrhage prediction in acute promyelocytic leukemia: validation of a risk score in a cohort from an international consortium treated with chemotherapy plus all-trans retinoic acid. Haematologica. 2025 Mar 1;110(3):795-798. doi: 10.3324/haematol.2024.286338. No abstract available. PMID 39479861
- [Background] Koury LCA, Kim HT, Undurraga MS, Navarro-Cabrera JR, Salinas V, Muxi P, Melo RAM, Gloria AB, Pagnano K, Nunes EC, Bittencourt RI, Rojas N, Quintana S, Ayala-Lugo A, Oliver AC, Figueiredo-Pontes L, Traina F, Moreira F, Fagundes EM, Duarte BKL, Mora-Alferez AP, Ortiz P, Untama J, Tallman M, Ribeiro R, Ganser A, Dillon R, Valk PJM, Sanz M, Lowenberg B, Berliner N, Rego EM. Clinical networking results in continuous improvement of the outcome of patients with acute promyelocytic leukemia. Blood. 2024 Sep 19;144(12):1257-1270. doi: 10.1182/blood.2024023890. PMID 38805638
- [Background] Correa de Araujo Koury L, Ganser A, Berliner N, Rego EM. Treating acute promyelocytic leukaemia in Latin America: lessons from the International Consortium on Acute Leukaemia experience. Br J Haematol. 2017 Jun;177(6):979-983. doi: 10.1111/bjh.14589. Epub 2017 May 3. PMID 28466545
- [Background] Rego EM, Kim HT, Ruiz-Arguelles GJ, Undurraga MS, Uriarte Mdel R, Jacomo RH, Gutierrez-Aguirre H, Melo RA, Bittencourt R, Pasquini R, Pagnano K, Fagundes EM, Chauffaille Mde L, Chiattone CS, Martinez L, Meillon LA, Gomez-Almaguer D, Kwaan HC, Garces-Eisele J, Gallagher R, Niemeyer CM, Schrier SL, Tallman M, Grimwade D, Ganser A, Berliner N, Ribeiro RC, Lo-Coco F, Lowenberg B, Sanz MA. Improving acute promyelocytic leukemia (APL) outcome in developing countries through networking, results of the International Consortium on APL. Blood. 2013 Mar 14;121(11):1935-43. doi: 10.1182/blood-2012-08-449918. Epub 2013 Jan 14. PMID 23319575